CLINICAL TRIAL: NCT02428595
Title: A Clinical Evaluation of the Eclipse™ System, a Vaginal Bowel Control (VBC) Therapy for Fecal Incontinence in Women
Acronym: LIBERATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pelvalon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA005
Record Dates: First submitted 2015-04-18; First posted 2015-04-29 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Eclipse™ System
  Interventions: Device: Eclipse™ System

INTERVENTIONS:
Device: Eclipse™ System — The Eclipse System is a vaginal bowel control (VBC) therapy intended to provide bowel control for women with fecal incontinence. It is comprised of a non-surgical device placed in the vagina (referred to as the "Eclipse Insert") and a pressure-regulated pump which is used to inflate and deflate the Insert. A Sizing Kit, for use during the fitting process, and an evaluation Insert (referred to as the Trial Insert) are also part of the Eclipse System.
  Other Names: Vaginal Bowel Control (VBC) Therapy

SUMMARY:
Multi-center, prospective, within-subject control, open label clinical trial to evaluate the durability of the safety and effectiveness of the Eclipse™ System after 3 and 12 months of use.

ELIGIBILITY:
Abbreviated Inclusion Criteria:

* History of Fecal Incontinence (FI) for at least 6 months
* Subject willing and able to give written informed consent to participate in the study
* Subject can read, write and communicate fluently in English
* Subject willing and able to comply with visit schedule
* Subject is able to physically manage the insertion and removal of the Insert

Abbreviated Exclusion Criteria:

* Vaginal childbirth within the last 18 months
* Currently pregnant or planning pregnancy during the study period
* Acute infections or genito-urinary injuries that would impact comfortable device use
* Current treatment for Fecal Incontinence other than medical management
* Removal or diversion of any portion of the bowel
* Recent urogenital or colorectal surgeries
* Chronic abdominal pain in absence of diarrhea
* Chronic (>6 mos) rectal, anal or pelvic pain
* Chronic watery diarrhea, unmanageable by drugs or diet
* Inflammatory Bowel Disease (IBD) such as Chron's or Ulcerative Colitis
* Rectal prolapse (mucosal or full thickness)
* Grade III or IV hemorrhoids
* Pelvic organ prolapse beyond the plane of the hymen
* Concurrent use of intra-vaginal pessary or other device
* Anal or pelvic malignancy within last 5 years
* History of pelvic irradiation for cancer
* Other significant medical or lifestyle factors that could confound the interpretation of the primary endpoint or increase subject risk

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Richter, PhD, MD, Principal Investigator — University of Alabama at Birmingham
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - University of North Carolina, Raleigh, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University (WIHRI), Providence, Rhode Island
  - Houston Methodist, Houston, Texas
  - Providence Sacred Heart, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Richter HE, Matthews CA, Muir T, Takase-Sanchez MM, Hale DS, Van Drie D, Varma MG. A vaginal bowel-control system for the treatment of fecal incontinence. Obstet Gynecol. 2015 Mar;125(3):540-547. doi: 10.1097/AOG.0000000000000639. PMID 25730213
- [Derived] Richter HE, Dunivan G, Brown HW, Andy U, Dyer KY, Rardin C, Muir T, McNevin S, Paquette I, Gutman RE, Quiroz L, Wu J. A 12-Month Clinical Durability of Effectiveness and Safety Evaluation of a Vaginal Bowel Control System for the Nonsurgical Treatment of Fecal Incontinence. Female Pelvic Med Reconstr Surg. 2019 Mar/Apr;25(2):113-119. doi: 10.1097/SPV.0000000000000681. PMID 30807411
- [Derived] Antosh DD, High R, Brown HW, Oliphant SS, Abed H, Philip N, Grimes CL. Feasibility of prophylactic salpingectomy during vaginal hysterectomy. Am J Obstet Gynecol. 2017 Nov;217(5):605.e1-605.e5. doi: 10.1016/j.ajog.2017.07.017. Epub 2017 Jul 20. PMID 28734829
- See also: A Vaginal Bowel-Control System for the Treatment of Fecal Incontinence (results of the LIFE Study) — http://journals.lww.com/greenjournal/Citation/2015/03000/A_Vaginal_Bowel_Control_System_for_the_Treatment.3.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients fit with the device, including patients that did not enter treatment. All subjects who completed the fitting process and entered the treatment period comprised the Intent-to-treat population. In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
Period: Fitting
Arm/Group | All Patients
Started | 137
Completed | 73
Not Completed | 64
Period: Treatment
Arm/Group | All Patients
Started | 73
Completed | 54
Not Completed | 19

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects who completed the fitting process and entered the treatment period comprised the Intent-to-treat population. In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
Arm/Group | All Subjects
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 51
  Black | 17
  Hispanic or Latino | 5
Region of Enrollment [Number; unit: participants]
  United States | 73
Body Mass Index [Number; unit: participants]
  <18.5 kg/m^2 | 1
  18.5 to <25 kg/m^2 | 23
  25 to <30 kg/m^2 | 27
  >=30 kg/m^2 | 22
Previous Gynecological Surgeries/Treatments [Count of Participants; unit: Participants]
  Hysterectomy | 30
  Prior prolapse surgery (excluding hysterectomy) | 10
  Prior urinary incontinence surgery | 10
  Gallbladder removal (Cholecystectomy) | 9
  Fistula repair | 1
  None of these | 28
Sexual Activity [Count of Participants; unit: Participants] | 37
Parity [Mean (Standard Deviation); unit: Pregnancies] | 2.2 (1.1)
Menopausal Status [Count of Participants; unit: Participants]
  Pre-menopause | 9
  Peri-menopause | 4
  Post-menopause | 60
Lower Urinary Tract and Bowel Conditions [Count of Participants; unit: Participants]
  Urinary incontinence | 22
  Overactive bladder (urinary frequency) | 34
  Irritable Bowel Syndrome (IBS) | 15
Duration of Fecal Incontinence Symptoms [Count of Participants; unit: Participants]
  6 months-5 years | 37
  >5 years | 36
Frequency of FI Symptoms (2 week period) [Mean (Standard Deviation); unit: count] | 14.1 (12.15)
Subjects with Fecal Urgency [Count of Participants; unit: Participants] | 53
Parity (Median) [Median (Full Range); unit: Pregnancies] | 2.0 [0 to 6]
Frequency of FI Symptoms (2 week period) (median) [Median (Full Range); unit: count] | 10.0 [4 to 83]

OUTCOME MEASURES:

1. Primary Outcome: Count of Treatment Responders in the Intent to Treat (ITT) Cohort
Description: Count of patients with >50% reduction in the average number of FI episodes per week as compared to baseline.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Intent to Treat: All subjects who completed the fitting process and entered the treatment period comprised the Intent-to-treat population. In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
Arm/Group | Intent to Treat
Number analyzed (Participants) | 73
Participants | 53

2. Secondary Outcome: Count of Treatment Responders in the Per Protocol (PP) Population
Description: Count of patients with >50% reduction in the average number of FI episodes per week as compared to Baseline.
Time Frame: 3, 6 and 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Per Protocol - 3 Months: Per Protocol cohort - 3 months is defined as all subjects who completed 3 months of the study without any major protocol deviations. In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
- Per Protocol - 6 Months: Per Protocol cohort - 6 months is defined as all subjects who completed 6 months of the study without any major protocol deviations. In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
- Per Protocol - 12 Months: Per Protocol cohort - 12 months is defined as all subjects who completed 12 months of the study without any major protocol deviations. In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
Arm/Group | Per Protocol - 3 Months | Per Protocol - 6 Months | Per Protocol - 12 Months
Number analyzed (Participants) | 63 | 57 | 54
Participants | 53 | 51 | 51

3. Secondary Outcome: Change in St. Mark's (Vaizey) Incontinence Severity Score as Compared to Baseline
Description: Change in mean scores on subject-reported outcomes related to symptom severity as reported by St. Mark's (Vaizey) Incontinence Severity Score.
  St. Mark's is a validated scale widely used in fecal incontinence research. The scale has a 24 point range where 0 = total fecal continence (better outcome) and 24 = total fecal incontinence (worse outcome). A reduction in the St. Mark's score is a better outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Per Protocol - 12 Months
Number analyzed (Participants) | 54
Score on a Scale | -6.9 (6.23)

4. Secondary Outcome: Change in Fecal Incontinence Quality of Life (FIQoL) Score as Compared to Baseline
Description: Change in mean score (from Baseline) on subject-reported outcomes as reported by FIQoL (Fecal Incontinence Quality of Life) score.
  The FIQoL scale asks a number of Fecal Incontinence (FI) related questions. Patient responses are rated from 1 to 4 points except one question which is rated from 1 to 5 points.
  The questions fall into four subscales: lifestyle, coping/behavior, depression/self-perception and embarrassment. The score for each subscale is the average of the responses in that group. For depression/self-perception the subscale score is from 1.0 to 5.0. The other subscale scores are from 1.0 to 4.0.
  The total FIQoL score is the sum of all four subscales, ranging from 4 to 17. For each subscale and the combined score, lower values indicate worse quality of life and higher values indicate better quality of life.
  An increase in score as compared to Baseline is therefore a better outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Per Protocol - 12 Months
Number analyzed (Participants) | 54
Score on a scale
  Change in Lifestyle Subscale score | 0.9 (0.79)
  Change in Coping/Behavior Subscale score | 1.1 (0.82)
  Change in Depression/Self Perception Subscalescore | 0.7 (0.75)
  Change in Embarrassment Subscale score | 1.2 (0.81)

5. Secondary Outcome: Numbers of Participants With Specific Patient Global Impression of Improvement (PGI-I) Scores
Description: The Patient Global Impression of Improvement (PGI-I) is a scale which describes the patient's perception of how their symptoms have change from Baseline.
  The scale has a range of 7 points from 1 to 7, where 1 = very much better than Baseline and 7 = very much worse than Baseline and 4 = no change from Baseline. A score below 4 is a better outcome and a score above 4 is a worse outcome, and a score of 4 is a neutral outcome.
  Note that because the patient is being asked to compare their symptoms to Baseline, no data is taken for this scale at Baseline and the score is an absolute value, not a change from a previous score.
Time Frame: 3, 6, 9 and 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Per Protocol - 9 Months: Per Protocol cohort - 9 months is defined as all subjects who completed 9 months of the study without any major protocol deviations. In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
- Per Protocol - 12 Months: Per Protocol cohort - 12 months is defined as all subjects who completed 12 months of the study without any major protocol deviations.
Arm/Group | Per Protocol - 3 Months | Per Protocol - 6 Months | Per Protocol - 9 Months | Per Protocol - 12 Months
Number analyzed (Participants) | 62 | 58 | 54 | 54
Participants
  Very Much Better | 26 | 26 | 29 | 29
  Much Better | 22 | 19 | 16 | 14
  A Little Better | 10 | 11 | 7 | 10
  No Change | 4 | 1 | 2 | 1
  A Little Worse | 0 | 1 | 0 | 0
  Much Worse | 0 | 0 | 0 | 0
  Very Much Worse | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: Safety Endpoint - Number of Device Related Adverse Events
Description: The number of device-related adverse events and device-related serious adverse events (related defined as probably or definitely).
  Events are classified as occurring either during fitting (the process of identifying the correct size of the device) or during treatment (defined as the time when a patient receives their long term wear device until the completion of the study).
Time Frame: 3, 6, 9 and 12 months
Measure: Number; unit: Count of Adverse Events
Groups:
- Treatment: All subjects who completed the fitting process and entered the treatment period comprised the Intent-to-treat population. In treatment, subjects wear the Eclipse Insert and inflate it 3x per day using the provided Pump. Patients can remove and reinsert the device as needed for cleaning or pelvic rest.
- Fitting: The period of time where a patient is fitted with the device in order to determine the correct size. All patients in the Treatment group are also present in the Fitting group. Adverse events which occurred in the Treatment phase are not included here.
Arm/Group | Treatment | Fitting
Number analyzed (Participants) | 73 | 137
Count of Adverse Events
  Non-serious adverse events (device related) | 44 | 90
  Serious adverse events (device related) | 0 | 0

ADVERSE EVENTS:
Time Frame: Events were collected for the full duration of study, including the fitting and treatment periods, for a total participation of 3.5-15 months (typically 13 months). For further detail, the fitting period, which occurs first, requires 2-4 weeks, but can be repeated up to 3 times, for a total of 2-12 weeks in this phase (typically 4 weeks). The treatment period, which follows the fitting period, is a minimum of 3 months and up to 12 months (typically 12 months).
Description: No difference in definitions. Adverse Event Categories: The majority of specific adverse events in this study occurred with very low frequency, which would not exceed common reporting thresholds. In order to provide a more accurate impression of the patient risk and to be more conservative in reporting, these low frequency events were gathered into groups by their systemic impact.
Groups:
- Fitting: All subjects who underwent the fitting process (interacted with a device), including those who did not enter the treatment period. The fitting process involved an office visit with a pelvic exam, followed by test fittings of the device to determine the correct size. Patients who were successfully fit then took home the Trial Insert device and wore it during the 2 weeks during which they collected diary data (logging bowel movements and incontinence episodes). This trial wear period was allowed to be extended due to scheduling or if the patient chose not to use the device during their menstrual cycle. Patients who did not achieve a successful fit were allowed to change device size and repeat the trial period up to 2 additional times (for a total of 3 fitting cycles).
- Treatment: All subjects who were successfully fit and completed their eligibility diary and who entered the 12 month treatment period. This includes patients who did not complete treatment. In treatment, subjects wore the Eclipse Insert and inflated it 3x per day using the provided Pump. Patients could remove and reinsert the device as needed for cleaning or pelvic rest.
Arm/Group | Fitting | Treatment
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/137 | 8/73
Other Adverse Events (participants affected / at risk) | 62/137 | 28/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fitting (N=137) | Treatment (N=73)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) — Not device related. Patient hospitalized for chest pain, underwent heart catheterization.
Suicidal ideations (Psychiatric disorders) | 0 (0) | 1 (1) — Not device related.
Breast cancer (Reproductive system and breast disorders) | 0 (0) | 2 (2) — Not device related.
Acute stroke (Nervous system disorders) | 0 (0) | 1 (1) — Not device related.
Chest discomfort (Cardiac disorders) | 0 (0) | 1 (1) — Not device related. Worsening dyspnea on exertion. Cardiac catheter and stent placement. History of coronary artery disease.
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not device related. History of interstitial lung disease.
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Not device related.
Worsening degenerative joint disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not device related. Worsening degenerative joint disease of bilateral hips.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fitting (N=137) | Treatment (N=73)
Vaginal Mucosal Wall Injury (Reproductive system and breast disorders) | 40 (46) | 10 (16) — Abrasion, bleeding, erythema, petechia, ecchymosis, hyperemia, or erosion of vaginal tissue apparent during pelvic examination.
Lower Urinary Tract Issues (Reproductive system and breast disorders) | 20 (21) | 7 (8) — New or increased urinary incontinence or voiding difficulty or urinary frequency, urinary tract infections, or dysuria.
Vaginal/Pelvic Discomfort/Irritation (Reproductive system and breast disorders) | 18 (20) | 11 (12) — Vaginal/Pelvic discomfort, pain, irritation, discharge, odor, burning sensation, or itching.
Vaginal Infections (Reproductive system and breast disorders) | 2 (2) | 5 (6) — Yeast infection of the vagina or unspecified vaginitis. Does not include systemic yeast infections or infections of other areas that do not affect the vagina.
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Leg pain.
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) — Constipation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT02428595/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT02428595/SAP_001.pdf